CLINICAL TRIAL: NCT01348581
Title: Chronic Wound Treatment With Extracellular Matrix (ECM) Scaffold Made From Fish Proteins
Brief Title: Use of Fish Skin Extracellular Matrix (ECM) to Facilitate Chronic Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KERECIS-10-106-S1; MW-ECM
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2011-05

CONDITIONS: Pressure Ulcers; Venous Ulcers; Diabetic Ulcers; Chronic Ulcer of Foot; Trauma-related Wound
Keywords: Adult; Aged; Aged, 80 and over; Bandages; Biological Dressings; Chronic Disease; Collagen; Epithelium; Extracellular Matrix; Fibroblasts; Granulation Tissue; Humans; Leg Ulcer; Middle Aged; Prospective Studies; Soft Tissue Injuries; Treatment Outcome; Varicose Ulcer; Wound Healing; Wounds and Injuries
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer; Chronic Disease; Leg Ulcer; Soft Tissue Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Marigen Wound Dressing (Experimental)
  Interventions: Device: Marigen Wound Dressing

INTERVENTIONS:
Device: Marigen Wound Dressing — The dressing is changed at least twice a week, with no more than five days between dressing changes. It is extremely important that the dressings are changed sufficiently often. On highly exuding ulcers the three or four dressing changes per week may be necessary. Duration is four weeks.

SUMMARY:
The clinical study is designed to assess the effectiveness, safety and non-immunogenicity of fish skin wound dressing extracellular matrix (ECM) in treating chronic wounds.

The wound dressing is indicated for the management of difficult to heal and chronic wounds. The matrix is cut to fit the wound and is applied to the wound bed. An absorptive secondary dressing is put on top. Further dressing of the wound depends on the etiology.

The indications for use are:

* partial and full-thickness wounds
* pressure ulcers
* venous ulcers
* diabetic ulcers
* chronic vascular ulcers
* tunneled/undermined wounds
* trauma wounds (abrasions, lacerations, second-degree burns, and skin tears)

ELIGIBILITY:
Inclusion Criteria:

* Venous leg ulcer
* Arterial leg ulcer
* Rheumatic leg ulcer
* Hydrostatic leg ulcer
* Ulcer where healing is delayed because of drug therapy
* Non-healing ulcer due to known or unknown causes

Exclusion Criteria:

* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | one year

SECONDARY OUTCOMES:
Wound granulation | one year

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Reykjavik, Iceland